CLINICAL TRIAL: NCT00573456
Title: Phase 1 Study to Evaluate the Efficacy of Using Energy Specific Far Infrared Radiation Treatment for Diabetes
Brief Title: Far Infrared Radiation Treatment for Diabetes
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GAAD Medical Research Institute Inc. (Other)
Responsible Party: Dr. Kwasi Donyina/Founder & President, GAAD Medical Research Institute Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAAD-DM-CTP1
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2009-08-17 (Estimated); Status verified 2009-08

CONDITIONS: Diabetes Mellitus
Keywords: Thye 1 Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other)
  Interventions: Radiation: Far Infrared Radiation

INTERVENTIONS:
Radiation: Far Infrared Radiation — Far Infrared Radiation (5μm to 20μm wavelength) for 30 to 40 minutes per session.

SUMMARY:
A study to determine the use of far infrared (FIR) radiation for treatment of diabetes.

DETAILED DESCRIPTION:
Diabetes mellitus is a disease in which glucose is not sufficiently metabolized. This results in high glucose levels in blood and glucose in the urine. Cells can starve because glucose is not being metabolized.

Both types of diabetes can cause dangerous complications, including blindness, heart and blood vessel disease, and kidney failure. A decrease in circulation may eventually require the amputation of limbs.

We are postulating that energy specific electromagnetic radiation of the central nervous system, the viscera and the endocrine system has the potential to enhance the immune system; thereby improving the health of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Persons with type 1 or type 2 diabetes

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-05; Primary Completion 2009-02 (Actual); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
The primary end point is to determine the therapeutic effects of far infrared radiation on all types of diabetes. | 2 years

SECONDARY OUTCOMES:
The secondary end point of the study is to evaluate the therapeutic effects of far infrared radiation on other types of diabetes complications including blindness, heart and blood vessel disease and kidney failure. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ken Nedd, M.D., Study Director — GAAD Medical Research Institute Inc.; Kwasi Donyina, Ph.D., Study Chair — GAAD Medical Research Institute Inc.
Locations (1):
- The Centre for Incurable Diseases, Toronto, Ontario, Canada